CLINICAL TRIAL: NCT02122705
Title: A Case Series of Vital Signs-controlled, Patient Assisted Intravenous Analgesia (VPIA) Using Remifentanil for Labour and Delivery
Brief Title: A Case Series of VPIA Using Remifentanil for Labour and Delivery
Acronym: VPIA
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIRB/2012/264/D
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2015-09

CONDITIONS: Labor Pain
Keywords: Remifentanil; Labour analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VPIA remifentanil: VPIA remifentanil labour analgesia
  Interventions: Device: VPIA remifentanil

INTERVENTIONS:
Device: VPIA remifentanil — Vital signs controlled patient assisted intravenous analgesia using remifentanil

SUMMARY:
This study is a prospective case series aiming to evaluate a new VPIA remifentanil algorithm which would benefit labouring mothers who are unable or unwilling to receive epidural analgesia.

DETAILED DESCRIPTION:
This study proposes a novel Vital signs-controlled, patient-assisted intravenous analgesia (VPIA) regimen that will enhance the efficacy, safety and personalization of remifentanil therapy for labouring women. This system will study the parturient's pattern of analgesic use in 15 min epochs and titrate the demand doses and basal infusion rate to maintain a plasma level of remifentanil that is appropriate for the degree of pain felt.

The system incorporates vital signs (pulse oximetry and heart rate values) into the algorithm which would temporarily stop the pumps and step down doses accordingly when predefined critical values are reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients who choose to use parenteral opioid for pain relief with informed consent
* Patients who refuse labour epidural analgesia
* Patients with contraindication to epidural analgesia (eg. Thrombocytopaenia, previous thoraco-lumbar spinal instrumentation)

Exclusion Criteria:

* Patients who are unable to understand instructions given regarding the use of patient controlled analgesia (PCA) or unable to self administer PCA boluses
* Patients with difficulty in communication due to language differences
* Patients with known hypersensitivity to remifentanil or any component of its formulation or to other fentanyl analogs
* Patients with severe respiratory disease
* Patients with history of drug dependence of recreational drug abuse
* Patients with unmanaged foetal bradycardia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Term parturients presenting to the hospital delivery suite in labour
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain score | Duration of labour
  Hourly maternal pain scores

SECONDARY OUTCOMES:
Remifentanil drug consumption | Duration of labour
  Total and hourly remifentanil drug consumption.
Maternal side effects | Duration of labour and 1st day post delivery
  Incidence of side effects : sedation, respiratory depression, oxygen desaturation, bradycardia, pruritus, nausea and vomiting
Maternal outcomes | Duration of labour and one day post delivery
  Mode of delivery Duration of second stage Overall satisfaction with labour analgesia

OTHER OUTCOMES:
Neonatal outcomes | Duration of labour and one day post delivery
  Birth weight APGAR scores at 1 and 5 minutes umbilical cord blood pH

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ling Leong, MBBS FANZCA, Principal Investigator — KK Women's & Children's Hospital
Locations (1):
- KK Women's & Children's Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No